CLINICAL TRIAL: NCT00141544
Title: A Multi-Center, Double-Blind Study to Determine the Efficacy of ESTRATEST® Tablets in Relieving Menopausal Symptoms in Estrogenized, Non-Hysterectomized Postmenopausal Women
Brief Title: The Efficacy of ESTRATEST® Tablets in Relieving Menopausal Symptoms in Estrogenized, Non-Hysterectomized Postmenopausal Women
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Cindy Lane, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S030.2.107
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Menopause
Keywords: Menopause; Postmenopause; Estrogen; Hormone Therapy
MeSH Terms: interventions — Estrogens, Esterified (USP); Methyltestosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: esterified estrogens 1.25 mg and methyltestosterone 2.5 mg
- 2 (Active Comparator)
  Interventions: Drug: Esterified estrogens 1.25 mg

INTERVENTIONS:
Drug: esterified estrogens 1.25 mg and methyltestosterone 2.5 mg — ESTRATEST® administered orally QD
  Arms: 1
Drug: Esterified estrogens 1.25 mg — Esterified estrogens 1.25 mg administered orally QD
  Arms: 2

SUMMARY:
To determine whether treatment with ESTRATEST® Tablets is superior to treatment with esterified estrogens tablets

ELIGIBILITY:
Inclusion Criteria:

Non-hysterectomized, menopausal women between the ages of 35 and 65 years (inclusive) with symptoms of estrogen and/or androgen deficiency not currently controlled by estrogen therapy as determined by patient report and the Investigator's clinical judgement

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-07; Primary Completion 2007-04 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total score of the Menopause Rating Scale (MRS) | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in the domain and individual item scores of the MRS | 12 weeks
Change from baseline in the domain scores of the MENQOL | monthly for 3 months
Comparison of changes in hormone levels and correlation with changes in the MRS | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (78):
- United States (78):
  - Site 66, Huntsville, Alabama
  - Site 57, Mobile, Alabama
  - Site 46, Montgomery, Alabama
  - Site 29, Phoenix, Arizona
  - Site 15, Tucson, Arizona
  - Site 3, Jonesboro, Arkansas
  - Site 22, Little Rock, Arkansas
  - Site 68, Carmichael, California
  - Site 55, Encinitas, California
  - Site 6, San Diego, California
  - Site 45, Santa Rosa, California
  - Site 25, Walnut Creek, California
  - Site 26, Denver, Colorado
  - Site 1, Groton, Connecticut
  - Site 54, Hartford, Connecticut
  - Site 30, Trumbull, Connecticut
  - Site 34, Waterbury, Connecticut
  - Site 10, Aventura, Florida
  - Site 78, Clearwater, Florida
  - Site 73, Fort Myers, Florida
  - Site 51, Leesburg, Florida
  - Site 49, Melbourne, Florida
  - Site 64, New Port Richey, Florida
  - Site 61, Ocala, Florida
  - Site 27, Palm Springs, Florida
  - Site 11, Pinellas Park, Florida
  - Site 75, Sarasota, Florida
  - Site 69, St. Petersburg, Florida
  - Site 70, Venice, Florida
  - Site 17, West Palm Beach, Florida
  - Site 50, Alpharetta, Georgia
  - Site 5, Atlanta, Georgia
  - Site 44, Decatur, Georgia
  - Site 77, Douglasville, Georgia
  - Site 9, Riverdale, Georgia
  - Site 7, Savannah, Georgia
  - Site 47, Boise, Idaho
  - Site 24, Champaign, Illinois
  - Site 20, Chicago, Illinois
  - Site 76, Peoria, Illinois
  - Site 58, Evansville, Indiana
  - Site 39, Wichita, Kansas
  - Site 59, Baton Rouge, Louisiana
  - Site 52, New Orleans, Louisiana
  - Site 53, Ann Arbor, Michigan
  - Site 63, Kansas City, Missouri
  - Site 32, Richmond Heights, Missouri
  - Site 36, St Louis, Missouri
  - Site 72, Billings, Montana
  - Site 21, Lincoln, Nebraska
  - Site 37, Reno, Nevada
  - Site 65, Cary, North Carolina
  - Site 13, New Bern, North Carolina
  - Site 16, Winston-Salem, North Carolina
  - Site 60, Columbus, Ohio
  - Site 67, Oklahoma City, Oklahoma
  - Site 40, Tulsa, Oklahoma
  - Site 62, Eugene, Oregon
  - Site 41, Medford, Oregon
  - Site 33, Portland, Oregon
  - Site 18, Erie, Pennsylvania
  - Site 19, Philadelphia, Pennsylvania
  - Site 23, Pottstown, Pennsylvania
  - Site 31, Anderson, South Carolina
  - Site 35, Greer, South Carolina
  - Site 4, Chattanooga, Tennessee
  - Site 74, Conroe, Texas
  - Site 8, Corpus Christi, Texas
  - Site 71, Dallas, Texas
  - Site 42, Houston, Texas
  - Site 14, San Antonio, Texas
  - Site 38, Salt Lake City, Utah
  - Site 28, Norfolk, Virginia
  - Site 12, Richmond, Virginia
  - Site 56, Renton, Washington
  - Site 2, Seattle, Washington
  - Site 48, Spokane, Washington
  - Site 43, Tacoma, Washington